CLINICAL TRIAL: NCT01798251
Title: A Randomized Single Center Phase II Study Comparing XELOX With Capecitabine Maintenance or XELOX Treatment in Elderly Metastatic Adenocarcinoma of Stomach
Brief Title: XELOX With Capecitabine Maintenance or XELOX in Elderly Metastatic Adenocarcinoma of Stomach
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Harbin Medical University (Other)
Responsible Party: Principal Investigator, BAI Yuxian, Professor, Harbin Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CGOG20120101009
Record Dates: First submitted 2012-12-13; First posted 2013-02-25 (Estimated); Last update posted 2013-05-06 (Estimated); Status verified 2013-05

CONDITIONS: Gastric Cancer
Keywords: Elderly Gastric Cancer; Capecitabine Maintenance
MeSH Terms: conditions — Stomach Neoplasms | interventions — Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- XELOX-X (Experimental): XELOX: Oxaliplatin: 100mg/m2 d1 Intravenous infusion, every 3 weeks. Capecitabine: 850mg/m^2 bid, days 1-14, every 3 weeks and maximum 4 cycles, or progression/intolerance.
  X Maintenance: Capecitabine 850mg/m^2 bid, days 1-14, every 3 weeks after 4 cycles XELOX regimen, until progression/intolerance.
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine
- XELOX (Active Comparator): XELOX: Oxaliplatin 100mg/m2 d1 Intravenous infusion, every 3 weeks. Capecitabine 850mg/m^2 bid, days 1-14, every 3 weeks, until progression/intolerance.
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine

INTERVENTIONS:
Drug: Oxaliplatin — Oxaliplatin 100mg/m2 d1 Intravenous infusion every 3 weeks
  Other Names: L-OHP
Drug: Capecitabine — capecitabine 850mg/m2 bid, d1-14, every 3 weeks
  Other Names: XELODA

SUMMARY:
To confirm the efficacy and safety of XELOX with capecitabine maintenance in treatment of elderly advanced gastric cancer (AGC) by comparing it with that of XELOX regimen.

DETAILED DESCRIPTION:
To investigate whether XELOX with capecitabine maintenance treatment as 1st line treatment in the elderly advanced gastric cancer is as effective and safe as XELOX regimen.

ELIGIBILITY:
Inclusion Criteria:

* Ages Eligible for Study: 65 Years or older
* Genders Eligible for Study: Both
* The Eastern Cooperative Oncology Group (ECOG) status ≤ 2
* Histologically confirmed gastric adenocarcinoma(including LAUREN type).
* Measurable disease(according to the Response Evaluation Criteria in Solid Tumors (RECIST) criteria 1.1).
* chemotherapy naive after recurrence or metastasis. Previous neo-adjuvant or adjuvant treatment for gastric cancer, if applicable, more than 6 months.
* Hb > 90g/L, neutrophil count > or = 1.5*10^9/L, platelet > or = 100*10^9/L, alanine transaminase (ALT) and aspartate aminotransferase (AST) < or = 2.5 times upper limit of nominal (ULN), alkaline phosphatase (ALP) < or = 2.5 times ULN, total bilirubin (TBIL) < 1.5 times ULN, serum albumin level > or = 30g/L, serum creatinine < 1 times ULN.
* No serious concomitant diseases which could lead to death within 5 years. At least 5 years from the last Biological/Immunotherapy/Hormone treatment for Malignancy excluding gastric cancer.
* Able to accept oral medication
* Compliance with protocol

Exclusion Criteria:

* Had received cytotoxic chemotherapy, radiotherapy or immunotherapy for this gastric cancer, excluding Corticosteroids.
* Other previous malignancy within 5 year, except curative skin cancer or carcinoma in situ of uterine cervix.
* Uncontrolled epilepsy, central nervous system disorders, or a history of mental disorders.
* clinically significant(i.e. active)cardiac disease e.g. symptomatic coronary artery disease, New York Heart Association (NYHA) II or more serious congestive heart failure or severe requiring medication intervention arrhythmia, or history of myocardial infarction within the last 12 months.
* Upper gastrointestinal obstruction or physiological dysfunction or suffering from malabsorption syndrome, which could affect the absorption of capecitabine.
* Organ transplantation requires immunosuppressive treatment.
* Severe uncontrolled recurrent infections, or Other serious uncontrolled concomitant diseases.
* Moderate or severe renal impairment(creatinine clearance (CCr) = or < 50 ml/min), or serum creatinine > ULN.
* Known enzyme deficiency of dihydropyrimidine dehydrogenase(DPD).
* Allergy to Oxaliplatin or any study medication ingredients.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-12; Primary Completion 2014-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months

SECONDARY OUTCOMES:
overall survival (OS) | from the date of randomization until death from any cause or up to 1 year
Response Rate (RR) | evaluate every 6 weeks after the date of randomization until diease progress or up to 12 weeks
adverse events (AE) | from date of randomization to 28 days after the last chemo dosage

OTHER OUTCOMES:
health-related quality of life (HRQOL) | evaluate every 6 weeks from the date of randomization until 28 days after the last chemo dosage
excision repair cross-complementing 1(ERCC1) expression | assays messager ribonucleic acid (mRNA) of ERCC1 expression in tumor tissue after randomization and before the first treatment
  quantitative real-time reverse transcriptase polymerase chain reaction (PCR) assays were performed to determine ERCC1 mRNA expression in tumor tissue.
K-ras gene type | assess after randomization and before the first treatment
  Genomic Deoxyribonucleic acid (DNA) is extracted from tumor tissue, direct sequencing technique is used to test K-ras gene type(mutation or wild).

CONTACTS AND LOCATIONS:
Overall Officials: Yuxian BAI, PhD, Principal Investigator — The tumor hospital of Harbin medical university
Locations (1):
- The tumor hospital of Harbin medical university, Harbin, Heilongjiang, China